CLINICAL TRIAL: NCT06436820
Title: The Relationship Between Intracranial Pressure and Aqueous Outflow in Idiopathic Intracranial Hypertension
Brief Title: ICP & Outflow Study
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 310393.
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Eye Change; Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected IIH patient group: Patients with suspected Idiopathic intracranial hypertension, who require a lumbar puncture as part of their standard care.
  Interventions: Procedure: Lumbar puncture
- Control group: Patients who require lumbar puncture for reasons not pertaining to raised intracranial pressure as part of their standard care.
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture — Lumbar puncture procedure performed within a clinical setting

SUMMARY:
This study aims to investigate the relationship between intracranial pressure (ICP) and aqueous outflow (the flow of the eye's internal fluid out of the eye), in patients with increased intracranial pressure (idiopathic intracranial hypertension (IIH)).

Through observing changes in aqueous outflow facility in patients scheduled for lumbar Puncture (LP) as part of their routine care the objectives we aim to answer include:

* Investigating the effect of lumbar puncture induced reduction in ICP on patients with known or suspected IIH, compared to control patients, who will be receiving LP for reasons not pertaining to high pressure.
* Comparing pre lumbar puncture aqueous outflow facility between patients with idiopathic intracranial hypertension and control patients.

Outside of the standard care provided for these patients as part of their scheduled lumbar puncture, they will have measurements of their eye taken before and after their lumbar puncture.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between intracranial pressure (ICP) and aqueous outflow (the flow of the eye's internal fluid out of the eye), in patients with increased intracranial pressure (idiopathic intracranial hypertension (IIH)).

The effect of lowering intracranial pressure on aqueous outflow will be examined by taking additional measurements before and after a procedure called a lumbar puncture (LP). These measurements include a scan to measure the dimensions of the eye, intraocular pressure reading, and a non-invasive technique to measure aqueous outflow (electronic Schiotz tonography) which is used regularly in the eye research unit at St Thomas' Hospital.

Study participants will already be scheduled for a lumbar puncture as they have known or suspected IIH, and LP is routinely used to investigate this. Additionally, control participants having LP for reasons not pertaining to a condition that may elevate intracranial pressure will also be included. Study participants will finish their involvement following the second aqueous outflow reading, after their LP.

A lumbar puncture procedure directly measures the intracranial pressure, but also reduces the pressure in the process. If aqueous outflow is measured before and after lumbar puncture, it will provide more information about whether the change in intracranial pressure affects the intraocular pressure due to a change in the rate of fluid flowing out of the eye. If a relationship between intracranial pressure and aqueous outflow is found to be present, it may offer an alternative non-invasive measurement for intracranial pressure. Additionally, this study would highlight an avenue of investigation into dysregulation of intraocular pressure in conditions such as glaucoma. Similarly, negative findings would help inform ongoing discussions and controversies in the literature regarding relationships between intraocular pressure and intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males or female between the ages of 18 and 80 (inclusive).
* Able to understand the study and give informed consent.
* Willing, able and available to participate in all aspects of the study.
* Able to undergo accurate tonography.
* Diagnosis of Idiopathic intracranial hypertension (IIH) or suspected diagnosis of IIH as determined by a consultant subspecialist neurologist or neuro-ophthalmologist.

Control group will only include:

* Individuals requiring lumbar puncture as part of their standard care for reasons other than suspected raised intracranial pressure e.g. for cerebrospinal fluid (CSF) sampling to analyse oligoclonal bands or other conditions necessitating lumbar puncture for diagnostic/prognostic purposes.
* Individuals suspected of having a raised intracranial pressure but, upon measurement of the opening pressure, are found to have an intracranial pressure within normal limits.*

  * In this study, where there are considered to be signs of raised intracranial pressure as judged by a consultant neuro ophthalmologist or neurologist, in combination with an opening CSF pressure 20cmH2O or greater, this will be taken as a raised intracranial pressure. Normal CSF pressure is taken as 19cmH2O or lower. In asymptomatic patients, pressures of up to 25cmH2O will be considered normal.

Exclusion Criteria

* Under 18 or over 80 years of age.
* Diagnosis of ocular hypertension (ocular hypertension is defined as any individual with an intraocular pressure above 24mmHg measured on Goldman tonometry, irrespective of corneal thickness. This applies to intraocular pressure measured historically as well on the day of assessment).
* Diagnosis of glaucoma of any subtype (glaucoma is defined on the basis of any glaucomatous optic nerve head appearance [including that defined on the basis of optic nerve head optical coherence tomography] or visual field defect, irrespective of intraocular pressure).
* Diagnosis of any significant retinal, corneal or other ocular abnormality aside from optic nerve head oedema secondary to raised ICP.
* Previous intraocular surgery or any surgery in which the conjunctiva has been breached e.g. optic nerve sheath fenestration or squint surgery.
* Diagnosis of raised intracranial pressure secondary to space occupying lesions.
* Any central nervous system or other systematic disorder that is likely to make lumbar puncture high risk or likely to render accurate recording of opening pressures unreliable.
* Mental impairment conflicting with informed consent.
* Patients who might not adequately understand written information given in English or verbal explanations in English will not be included as participants in the study must be able to understand English to complete some of the tests.
* Participants will not be included if they are involved in research deemed by the investigators to impact the outcomes of this study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from neuro-ophthalmology clinics and neurology clinics in St Thomas hospital London UK
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Measure the effect of LP induced change in intracranial pressure on outflow facility in patients with idiopathic intracranial hypertension compared to control patients | 18 Months
  To investigate the effect of lumbar puncture induced changes in intracranial pressure on aqueous outflow facility in patients with known or suspected idiopathic intracranial hypertension, compared to control patients.

SECONDARY OUTCOMES:
Measure the difference in outflow facility between patients with idiopathic intracranial hypertension and control patients prior to lumbar puncture | 18 Months
  To compare pre lumbar puncture aqueous outflow facility between patients with idiopathic intracranial hypertension and control patients.

IPD SHARING:
Plan to Share IPD: No